CLINICAL TRIAL: NCT05229835
Title: Effect of Time-restricted Eating and Endurance Training on Markers of the Health of Women and Men-role of Dietary Supplements
Brief Title: Effect of Time-restricted Eating and Endurance Training on Markers of the Health of Women and Men
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 04-0246/09/306
Record Dates: First submitted 2022-01-14; First posted 2022-02-08 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Physical Exercise; Time Restricted Eating; Mental Health Wellness 1; Wellbeing; Biochemical Markers
Keywords: time restricted eating; exercise; supplementation; iron; oxidative stress
MeSH Terms: conditions — Motor Activity; Intermittent Fasting | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Intervention studies
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Time restricted eating (Experimental): Tasks for participants are to fast for 14 h during the day and eat 10h during 12 weeks period
  Interventions: Other: Time restricted eating and exercise
- Time restricted eating combined with exercise (Experimental): Tasks for participants are to fast for 14 h during the day and eat 10h during 12 weeks period combined with aerobic exercise 3 times a week.
  Interventions: Other: Time restricted eating and exercise
- Exercise (Experimental): Tasks for participants are to perform aerobic exercise 3 times a week.
  Interventions: Other: Time restricted eating and exercise
- Control (No Intervention): Tasks for participants are keeping their daily habits

INTERVENTIONS:
Other: Time restricted eating and exercise — We apply time restricted eating, exercise alone and combined
  Arms: Exercise; Time restricted eating; Time restricted eating combined with exercise

SUMMARY:
The aim of this project is to demonstrate the synergistic effect of TRE and NW training on health indicators for older women. The women will be divided into four groups, i.e. Control group (CG); time-restricted eating group (TRG) which will follow 12 weeks of TRE protocol; Nordic walking training group (NWT) which will follow 12 weeks of supervised Nordic walking training and Nordic walking training combined with a time-restricted eating group (NW-TRG). In addition, it is assumed to prove that among young men, TRE will improve adaptation to endurance training and improve the metabolism. The study will be divided into two groups: 1. a group undergoing endurance training and 2. a group combining endurance training with TRE. In all subject's changes in the metabolism of iron, tryptophan, vitamin D and lipids will be evaluated. Endocrine function of skeletal muscles, mental state and cognitive abilities of the subjects will also be examined. The investigators expect that the applied procedure of temporary restriction of food intake will be easy to apply and continue for much longer than the study period. In order to maintain this time window, test subjects will be asked to delay their breakfast and early dinner intake. In addition, it is expected that the improvement in wellbeing, vitality and a significant improvement in performance and biochemical indicators of health, especially in the NWT plus TRE group, will allow to better understand the physiology of exercise, which may result in future specific health recommendations for people of different ages.

DETAILED DESCRIPTION:
Studies of recent years prove that one of the important causes of metabolic disorders in people is a disturbed daily cycle, which is significantly influenced by the time of eating. It has been shown that more than 50% of the examined persons consumed food for 15 hours and more during the day. Limiting food consumption to 8-10 hours, without the need to reduce food intake, the so-called time-restricted eating (TRE), resulted in a significant improvement in metabolism, decrease in body weight and cholesterol concentration, increase in insulin sensitivity and many others. A period of hunger is necessary for the body to regenerate cell structures and allows for the separation of opposing metabolic processes. This means that the period of hunger is necessary and its limitation by e.g. snacking can seriously disturb this series of processes in the human body. The results of the investigators preliminary research indicate that TRE increases the vitality of the examined persons and their desire for doing exercise. So far, there are no studies on older people, where the intervention would consist in the use of TRE and endurance training such as Nordic walking (NW). The aim of this project is to demonstrate the synergistic effect of TRE and NW training on health indicators for older women. The women will be divided into four groups, i.e. Control group (CG); time-restricted eating group (TRG) which will follow 12 weeks of TRE protocol; Nordic walking training group (NWT) which will follow 12 weeks of supervised Nordic walking training and Nordic walking training combined with a time-restricted eating group (NW-TRG). In addition, it is assumed to prove that among young men, TRE will improve adaptation to endurance training and improve the metabolism. The study will be divided into two groups: 1. a group undergoing endurance training and 2. a group combining endurance training with TRE. In all subject's changes in the metabolism of iron, tryptophan, vitamin D and lipids will be evaluated. Endocrine function of skeletal muscles, mental state and cognitive abilities of the subjects will also be examined. The investigators expect that the applied procedure of temporary restriction of food intake will be easy to apply and continue for much longer than the study period. In order to maintain this time window, test subjects will be asked to delay their breakfast and early dinner intake. In addition, it is expected that the improvement in wellbeing, vitality and a significant improvement in performance and biochemical indicators of health, especially in the NWT plus TRE group, will allow to better understand the physiology of exercise, which may result in future specific health recommendations for people of different ages.

ELIGIBILITY:
Inclusion Criteria:

* medical checkup
* good health status

Exclusion Criteria:

* acute cardiovascular disease
* acute respiratory disease
* stable hypertension,
* blood pressure over 160/100 mmHg
* pregnancy

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Time restricted eating and physical performance | 12 weeks
  The impact of this procedure on physical performance
Time restricted eating and mental performance | 12 weeks
  The impact of this procedure on mental performance
Time restricted eating and iron metabolism | 12 weeks
  The impact of this procedure on iron metabolism
Time restricted eating and myokines concentration | 12 weeks
  The impact of this procedure on myokinins concentration
Time restricted eating and lipid metabolism | 12 weeks
  The impact of this procedure on lipid metabolism
Time restricted eating and glucose metabolism | 12 weeks
  The impact of this procedure on glucose metabolism
Time restricted eating and tryptophan metabolism | 12 weeks
  The impact of this procedure on tryptophan metabolism
Time restricted eating and vitamin D metabolism | 12 weeks
  The impact of this procedure on vitamin D metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Jędrzej Antosiewicz, Ph.D., Principal Investigator — Medical University of Gdansk
Locations (1):
- Medical University of Gdańsk Faculty of Health Science, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kortas JA, Reczkowicz J, Juhas U, Ziemann E, Swiatczak A, Prusik K, Olszewski S, Soltani N, Rodziewicz-Flis E, Flis D, Zychowska M, Galezowska G, Antosiewicz J. Iron status determined changes in health measures induced by nordic walking with time-restricted eating in older adults- a randomised trial. BMC Geriatr. 2024 Mar 29;24(1):300. doi: 10.1186/s12877-024-04876-8. PMID 38553690